CLINICAL TRIAL: NCT05947240
Title: Effects of Upper Extremity Aerobic Exercise on Exercise Capacity and Physical Activity in Patients With Pulmonary Arterial Hypertension.
Brief Title: Effects of UE Aerobic Exercise on Exercise Capacity and PA in Patients With Pulmonary Arterial Hypertension.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0322
Record Dates: First submitted 2023-06-14; First posted 2023-07-17 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: Upper Extremity Aerobic Exercise Training;; ; Exercise Capacity; Rehabilitation
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Group A will be training group and group B will be control group. Deep breathing exercises will be done as baseline treatment in both groups. Both groups will be assessed with Modified Borg scale, 6-PBRT and Fatigue severity scale at the baseline. The control group patients will perform functional active alternating movements for the upper limbs at home involving three sets with 10 repetitions and a rest interval between 1- and 2-minute.
  Intervention will be for 3 times a week or 6 weeks
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- upper extremity aerobic exercises (Experimental): The treatment group patients will perform upper extremity aerobic exercises by using an arm ergometer under the supervision of a physiotherapist. Training intensity will adjust according to 50 80 % of max HR or intensity of dyspnea to 4 points on modified Borg scale (MBS) for at least 15 45 min,3 times/week over 6 weeks.
  Interventions: Other: aerobic exercises
- active alternating movements for the upper limbs a (Experimental): The control group patients will perform functional active alternating movements for the upper limbs at home involving three sets with 10 repetitions and a rest interval between 1- and 2-minute. Intervention will be for 3 times a week or 6 weeks.
  Interventions: Other: active alternating movements for the upper limbs

INTERVENTIONS:
Other: aerobic exercises — The treatment group patients will perform upper extremity aerobic exercises by using an arm ergometer under the supervision of a physiotherapist.
  Arms: upper extremity aerobic exercises
Other: active alternating movements for the upper limbs — The control group patients will perform functional active alternating movements for the upper limbs at home involving three sets with 10 repetitions and a rest interval between 1- and 2-minute. Intervention will be for 3 times a week or 6 weeks.
  Arms: active alternating movements for the upper limbs a

SUMMARY:
Group A will be training group and group B will be control group. Deep breathing exercises will be done as baseline treatment in both groups. Both groups will be assessed with Modified Borg scale, 6-PBRT and Fatigue severity scale at the baseline. The control group patients will perform functional active alternating movements for the upper limbs at home involving three sets with 10 repetitions and a rest interval between 1- and 2-minute.

Intervention will be for 3 times a week or 6 weeks. The treatment group patients will perform upper extremity aerobic exercises by using an arm ergometer under the supervision of a physiotherapist. Training intensity will adjust according to 50 80 % of max HR or intensity of dyspnea to 4 points on modified Borg scale (MBS) for at least 15 45 min, 3 times/week over 6 weeks.

DETAILED DESCRIPTION:
Group A will be training group and group B will be control group. Deep breathing exercises will be done as baseline treatment in both groups. Both groups will be assessed with Modified Borg scale, 6-PBRT and Fatigue severity scale at the baseline. The control group patients will perform functional active alternating movements for the upper limbs at home involving three sets with 10 repetitions and a rest interval between 1- and 2-minute.

Intervention will be for 3 times a week or 6 weeks. The treatment group patients will perform upper extremity aerobic exercises by using an arm ergometer under the supervision of a physiotherapist. Training intensity will adjust according to 50 80 % of max HR or intensity of dyspnea to 4 points on modified Borg scale (MBS) for at least 15 45 min, 3 times/week over 6 weeks. This study will measure and record HR by using the heart rate monitor, oxygen saturation (SpO2) by using pulse oximetry and blood pressure, breathing frequency (BF), dyspnea, fatigue, and arm fatigue by using MBS before, during, and after training.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with pulmonary arterial hypertension.
* Both the sex was considered.
* Age range from 35 to 60 years.
* Patients who were stable.
* Patient under optimal medical therapy for at least three months before participating in this study
* Willing to participate in study (13).

Exclusion Criteria:

* Patient with cognitive disorders.
* Patient with orthopedic or neurological diseases. acute infection or pneumonia
* Patient with class IV heart failure.
* Patient with acute infection or pneumonia.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
6 MWT | 4 weeks
  The 6MWT is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD).The self-paced 6MWT assesses the submaximal level of functional capacity.
Borg rating of perceived exertion (RPE) | 4 weeks
  Borg rating of perceived exertion (RPE) is an outcome measure scale used in knowing exercise intensity prescription. It is used in monitoring progress and mode of exercise in cardiac patients as well as in other patient populations undergoing rehabilitation and endurance training.Borg RPE scale was developed by Gunnar Borg for rating exertion and breathlessness during physical activity ; that is, how hard the activity is as shown by high heart and respiration rate , profuse perspiration and muscle exertion.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, MS.CPPT, Principal Investigator — Riphah International University
Locations (1):
- National hospital and Ittefaq hospital in Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malenfant S, Lebret M, Breton-Gagnon E, Potus F, Paulin R, Bonnet S, Provencher S. Exercise intolerance in pulmonary arterial hypertension: insight into central and peripheral pathophysiological mechanisms. Eur Respir Rev. 2021 Apr 13;30(160):200284. doi: 10.1183/16000617.0284-2020. Print 2021 Jun 30. PMID 33853885
- [Background] Karapolat H, Cinar ME, Tanigor G, Nalbantgil S, Kayikcioglu M, Mogulkoc N, Kultursay H. Effects of cardiopulmonary rehabilitation on pulmonary arterial hypertension: A prospective, randomized study. Turk J Phys Med Rehabil. 2019 May 8;65(3):278-286. doi: 10.5606/tftrd.2019.2758. eCollection 2019 Sep. PMID 31663077
- [Background] Cedeno de Jesus S, Almadana Pacheco V, Valido Morales A, Muniz Rodriguez AM, Ayerbe Garcia R, Arnedillo-Munoz A. Exercise Capacity and Physical Activity in Non-Cystic Fibrosis Bronchiectasis after a Pulmonary Rehabilitation Home-Based Programme: A Randomised Controlled Trial. Int J Environ Res Public Health. 2022 Sep 3;19(17):11039. doi: 10.3390/ijerph191711039. PMID 36078768
- [Background] Waller L, Kruger K, Conrad K, Weiss A, Alack K. Effects of Different Types of Exercise Training on Pulmonary Arterial Hypertension: A Systematic Review. J Clin Med. 2020 Jun 2;9(6):1689. doi: 10.3390/jcm9061689. PMID 32498263
- [Background] McCormack C, Kehoe B, Hardcastle SJ, McCaffrey N, McCarren A, Gaine S, McCullagh B, Moyna N. Pulmonary hypertension and home-based (PHAHB) exercise intervention: protocol for a feasibility study. BMJ Open. 2021 May 10;11(5):e045460. doi: 10.1136/bmjopen-2020-045460. PMID 33972341
- [Background] Zeng X, Chen H, Ruan H, Ye X, Li J, Hong C. Effectiveness and safety of exercise training and rehabilitation in pulmonary hypertension: a systematic review and meta-analysis. J Thorac Dis. 2020 May;12(5):2691-2705. doi: 10.21037/jtd.2020.03.69. PMID 32642177